CLINICAL TRIAL: NCT02513004
Title: Evaluation of Antiplatelet Effects and Safety of Intraoperative Administration of Ticagrelor Versus Clopidogrel in Patients Undergoing "One-stop" Hybrid Coronary Revascularization
Brief Title: Evaluation of Antiplatelet Effects and Safety of Intraoperative Administration of Ticagrelor Versus Clopidogrel
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yongjian Wu (Other)
Responsible Party: Sponsor-Investigator, Yongjian Wu, Professor, Chinese Academy of Medical Sciences, Fuwai Hospital
Organization: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-ZX46
Record Dates: First submitted 2015-06-14; First posted 2015-07-31 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor (Experimental): Patients will receive first dose of 90mg ticagrelor tablets (powdered) taken via nasogastric tube after LIMA-LAD bypass establishing, the close of thorax and before PCI procedure, followed by 90mg of ticagrelor 12 hours after the first dose.Thereafter, the patients will take 90mg of ticagrelor orally bid, at approximately 12-hourly intervals. The total study period is 3 months.
  Interventions: Drug: Ticagrelor
- Clopidogrel (Active Comparator): Patients will receive a loading dose of 300mg clopidogrel tablets (four 75mg capsules powdered) taken via nasogastric tube after LIMA-LAD bypass establishing, the close of thorax and before PCI procedure. Thereafter, the patients will take 75mg of clopidogrel capsules orally od. The total study period is 3 months.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — Patients will receive first dose of 90mg ticagrelor tablets (powdered) taken via nasogastric tube after LIMA-LAD bypass establishing, the close of thorax and before PCI procedure, followed by 90mg of ticagrelor 12 hours after the first dose. The third dose of ticagrelor will be given to patients after the 24 hour blood sample has been obtained and 24 hours after the first dose. Thereafter, the patients will take 90mg of ticagrelor orally bid, at approximately 12-hourly intervals. The total study period is 3 months.
  Other Names: BRILINTA
  Arms: Ticagrelor
Drug: Clopidogrel — Patients will receive a loading dose of 300mg clopidogrel tablets (four 75mg capsules powdered) taken via nasogastric tube after LIMA-LAD bypass establishing, the close of thorax and before PCI procedure. The second dose of clopidogrel will be given to patients after the 24 hour blood sample has been obtained and 24 hours after the first dose. Thereafter, the patients will take 75mg of clopidogrel capsules orally od. The total study period is 3 months.
  Other Names: PLAVIX
  Arms: Clopidogrel

SUMMARY:
This study is designed to test the hypothesis that the onset of the antiplatelet effect 90mg-first-dose of ticagrelor will be more rapid and greater than 300mg-loading-dose of clopidogrel evaluated by P2Y12 reaction units measured by Verify NowTM P2Y12 assay at 1 hour in patients undergoing one-stop Hybrid coronary revascularization(HCR).

DETAILED DESCRIPTION:
This is a single-center, randomized, active-controlled, open-label, prospective study, and the study is designed to test the hypothesis that the onset of the antiplatelet effect 90mg-first-dose of ticagrelor will be more rapid and greater than 300mg-loading-dose of clopidogrel evaluated by P2Y12 reaction units (PRU) measured by Verify NowTM P2Y12 assay at 1 hour in patients undergoing one-stop HCR. The first dose of study drug (ticagrelor 90mg or clopidogrel 300 mg) will be administered as powder via a nasogastric tube after conﬁrmation of left internal mammal artery to left anterior descending coronary antery (LIMA-LAD) graft patency during the HCR procedure. Approximately 60 patients will enrol for the study. Patients will be randomized equally (ratio 1:1) to the two treatment arms of this study. The anticipated duration of the study is approximately 15 months, including an anticipated enrolment period of 12 months and follow-up period of 3months.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. A patient who is considered as ethnic Chinese
3. 80years >aged> 18years, male or female
4. Patient is willing to perform HCR with the following conditions: Multi-vessel coronary artery disease with unfavorable left anterior descending coronary artery (LAD) for percutaneous coronary intervetion (PCI) (i.e., chronic total occlusion, excessive tortuosity, severely diffuse lesion), unprotected left main coronary artery disease, and non-LAD lesions were technically feasible for PCI with a drug-eluting stent (DES) .Limitations to traditional coronary artery bypass graft (CABG), such as pre-existing organ dysfunction, heavily calciﬁed proximal aorta, or lack of suitable graft conduits

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study
2. Previous enrolment or randomization in the present study
3. Participation in another clinical study with an investigational product during the last 30 days
4. Contraindication or other reason that clopidogrel or ticagrelor should not be administered (eg, hypersensitivity, active bleeding, moderate or severe liver disease, history of previous intracranial bleed, GI bleed within the past 6 months, major surgery within 30 days)
5. With coagulation disorder
6. With uric acid nephropathy
7. History of intolerance or allergy to acetylsalicylic acid (ASA) or clopidogrel or ticagrelor
8. Patient has a coronary artery bypass graft (CABG) history.
9. left subclavian artery and LIMA stenosis
10. buried intramyocardial LAD
11. need for a concomitant operation (e.g., valve repair or replacement)
12. overt congestive heart failure
13. Unsuccessful LIMA-LAD graft
14. hemodynamic instability
15. other conditions rendering PCI unsuitable (e.g., fresh thrombus, coronary vessel diameter <1.5 mm)
16. Platelet count less than 100*10^9/L
17. Haemoglobin (Hb) level less than 110g/L
18. White blood cell count less than 4*10^12/L
19. Recent (within 30 days of dosing) blood donation
20. Fibrinolytic therapy in the 24 hours prior to randomisation, or planned fibrinolytic treatment following randomisation (eg, for ST-segment elevation myocardial infarction or pulmonary embolism)
21. P2Y12 receptor inhibitor therapy in 7 days before HCR surgery.
22. Nonselective non-steroidal anti-inflammatory drugs (NSAIDs) and prostacyclins (PGI2) therapy that cannot be stopped
23. Increased risk of bradycardic events (eg, no pacemaker and known sick sinus syndrome, second degree atrioventricular block, third degree atrioventricular block or previous documented syncope suspected to be due to bradycardia).
24. Concomitant oral or intravenous therapy (see examples below) with strong CYP3A inhibitors, CYP3A substrates with narrow therapeutic indices, or strong CYP3A inducers within 14 days of study treatment or cannot be stopped for the course of the study.

    Strong inhibitors: ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, nefazadone, ritonavir, saquinavir, nelfinavir, indinavir, atanazavir, over 1 litre daily of grapefruit juice.

    Substrates with narrow therapeutic index: cyclosporine, quinidine. Strong inducers: rifampin/rifampicin, phenytoin, carbamazepine. The sponsor should be consulted for enrolment with any concomitant medicines which are suspected of undergoing strong drug-drug interaction
25. Any other condition which in the opinion of the investigator, may either put the patient at risk or influence the result of the study (e.g., cardiogenic shock or active cancer)
26. Moderate or severe renal disease;
27. Moderate or severe chronic lung disease or asthma;
28. Pregnancy or lactation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-03 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
1hourPRU | 1hour
  PRU measured by Verify NowTM P2Y12 assay at 1 hour after first dose of study drug administered as powder via a nasogastric tube after conﬁrmation of LIMA-LAD graft patency during the HCR procedure in HCR patients.

SECONDARY OUTCOMES:
30min,1h,2h,6h,12h,24h PRU | 30min,1h,2h,6h,12h,24h after first dose
  PRU measured by Verify NowTM P2Y12 assay at 30min,1h, 2h，6h,12h,24h after first dose of study drugs.

OTHER OUTCOMES:
safety assessed by the bleeding risk of ticagrelor compared with clopidogrel in the peri-operative and in-hospital period and 3 months follow-up. | 3 monthes

CONTACTS AND LOCATIONS:
Overall Officials: Yongjian Wu, Professor, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Shen L, Hu S, Wang H, Xiong H, Zheng Z, Li L, Xu B, Yan H, Gao R. One-stop hybrid coronary revascularization versus coronary artery bypass grafting and percutaneous coronary intervention for the treatment of multivessel coronary artery disease: 3-year follow-up results from a single institution. J Am Coll Cardiol. 2013 Jun 25;61(25):2525-33. doi: 10.1016/j.jacc.2013.04.007. Epub 2013 Apr 23. PMID 23623906
- [Result] Hu S, Li Q, Gao P, Xiong H, Zheng Z, Li L, Xu B, Gao R. Simultaneous hybrid revascularization versus off-pump coronary artery bypass for multivessel coronary artery disease. Ann Thorac Surg. 2011 Feb;91(2):432-8. doi: 10.1016/j.athoracsur.2010.10.020. PMID 21256284
- [Result] Wallentin L, Becker RC, Budaj A, Cannon CP, Emanuelsson H, Held C, Horrow J, Husted S, James S, Katus H, Mahaffey KW, Scirica BM, Skene A, Steg PG, Storey RF, Harrington RA; PLATO Investigators; Freij A, Thorsen M. Ticagrelor versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2009 Sep 10;361(11):1045-57. doi: 10.1056/NEJMoa0904327. Epub 2009 Aug 30. PMID 19717846
- [Result] Eikelboom JW, Hirsh J, Spencer FA, Baglin TP, Weitz JI. Antiplatelet drugs: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e89S-e119S. doi: 10.1378/chest.11-2293. PMID 22315278
- [Result] Kuliczkowski W, Witkowski A, Polonski L, Watala C, Filipiak K, Budaj A, Golanski J, Sitkiewicz D, Pregowski J, Gorski J, Zembala M, Opolski G, Huber K, Arnesen H, Kristensen SD, De Caterina R. Interindividual variability in the response to oral antiplatelet drugs: a position paper of the Working Group on antiplatelet drugs resistance appointed by the Section of Cardiovascular Interventions of the Polish Cardiac Society, endorsed by the Working Group on Thrombosis of the European Society of Cardiology. Eur Heart J. 2009 Feb;30(4):426-35. doi: 10.1093/eurheartj/ehn562. Epub 2009 Jan 27. PMID 19174428
- [Result] Gurbel PA, Bliden KP, Zaman KA, Yoho JA, Hayes KM, Tantry US. Clopidogrel loading with eptifibatide to arrest the reactivity of platelets: results of the Clopidogrel Loading With Eptifibatide to Arrest the Reactivity of Platelets (CLEAR PLATELETS) study. Circulation. 2005 Mar 8;111(9):1153-9. doi: 10.1161/01.CIR.0000157138.02645.11. Epub 2005 Feb 28. PMID 15738352
- [Result] Gurbel PA, Bliden KP, Butler K, Tantry US, Gesheff T, Wei C, Teng R, Antonino MJ, Patil SB, Karunakaran A, Kereiakes DJ, Parris C, Purdy D, Wilson V, Ledley GS, Storey RF. Randomized double-blind assessment of the ONSET and OFFSET of the antiplatelet effects of ticagrelor versus clopidogrel in patients with stable coronary artery disease: the ONSET/OFFSET study. Circulation. 2009 Dec 22;120(25):2577-85. doi: 10.1161/CIRCULATIONAHA.109.912550. Epub 2009 Nov 18. PMID 19923168
- [Result] Li Y, Zheng Z, Xu B, Zhang S, Li W, Gao R, Hu S. Comparison of drug-eluting stents and coronary artery bypass surgery for the treatment of multivessel coronary disease: three-year follow-up results from a single institution. Circulation. 2009 Apr 21;119(15):2040-50. doi: 10.1161/CIRCULATIONAHA.108.819730. Epub 2009 Apr 6. PMID 19349321
- [Result] Vandvik PO, Lincoff AM, Gore JM, Gutterman DD, Sonnenberg FA, Alonso-Coello P, Akl EA, Lansberg MG, Guyatt GH, Spencer FA. Primary and secondary prevention of cardiovascular disease: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e637S-e668S. doi: 10.1378/chest.11-2306. PMID 22315274